CLINICAL TRIAL: NCT06001281
Title: Predictive Value of Soluble CD146 in Patients With Recurrent Glioblastoma Treated by Bevacizumab
Brief Title: Predictive Value of Soluble CD146 in Glioblastoma Patients
Acronym: MUCIGLIO-01
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RCAPHM23_0011; ID RCB (Other: 2023-A00536-39)
Record Dates: First submitted 2023-08-14; First posted 2023-08-21 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2023-08

CONDITIONS: Glioblastoma
Keywords: glioblastoma; CD146; bevacizumab
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- plasma collection (Other): Plasma samples will be prospectively collected at relevant time points during patient treatment.
  Interventions: Other: plasma collection

INTERVENTIONS:
Other: plasma collection — Plasma samples will be prospectively collected at relevant time points during patient treatment.

SUMMARY:
Glioblastoma is the most common malignant primary brain tumor with poor prognosis because of its diffusive and infiltrative nature. The FDA approved the use of the anti-VEGF antibody bevacizumab in recurrent GBM. However, resistance to this anti-angiogenic reagent is frequent and fails to enhance patients' overall survival. The investigators previously identified one novel mechanism responsible for bevacizumab-resistance in CD146-positive glioblastoma (Joshkon et al. Acta Neuropathol Commun, 2022).

Now, the investigators objective is to prospectively monitor the soluble CD146 value in plasma from patients treated by bevacizumab for recurrent glioblastoma.

The investigators will collect plasma at baseline, before the first bevacizumab administration, before the second administration, at the time of first MRI evaluation and at progression. Plasma CD146 value will be analyzed by ELISA.

The investigators expect to confirm the correlation between soluble CD146 value in plasma and patient response to bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

* - Adult patients with recurrent IDHwt glioblastoma
* Relapse after standard first line treatment (radio-chemotherapy)
* Candidate for bevacizumab treatment
* Able to be monitored by MRI
* KPS ≥ 60%
* Written signed consent form

Exclusion Criteria:

* Pregnancy or breast feeding
* Life expectancy less than 3 months
* Bevacizumab in first line treatment
* Other concomitant life-threatening disease
* Under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2024-01-30 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
correlation between soluble CD146 plasma value and patient response (RANO) | first evaluation (2 months)
  Soluble CD146 plasma value will be assessed using ELISA. Patient response will be evaluated by MRI and clinical response using the international RANO criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Emeline Tabouret, Principal Investigator — AP-HM
Locations (1):
- Service de Neuro-oncologie, Marseille, France

IPD SHARING:
Plan to Share IPD: No